CLINICAL TRIAL: NCT05182216
Title: Social Media Use in Sickle Cell Patients
Status: Withdrawn | Type: Observational
Why Stopped: We have withdrawn this study.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sonja Smith, Program Manager, University of Alabama at Birmingham
Other Study IDs: 300007766
Record Dates: First submitted 2021-11-22; First posted 2022-01-10 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Survey, Family Life

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surveys of patients to identify primary social media sources for health news.

ELIGIBILITY:
Inclusion Criteria:

* sickle cell disease diagnosis

Exclusion Criteria:

* negative sickle cell disease diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with diagnosis of sickle cell disease
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Social Media Use in Sickle Cell Patients | six months
  Surveys. The survey will have a variety of social media options and ask participants to select the medium used to receive information on health, news, and entertainment.